CLINICAL TRIAL: NCT04224233
Title: iLiFE: a Home-based Physical Activity Programme for Patients With Advanced Interstitial Lung Diseases
Brief Title: A Home-based Physical Activity Programme for Patients With Advanced Interstitial Lung Diseases (iLiFE)
Acronym: iLiFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Centro Hospitalar do Baixo Vouga (Other)
Responsible Party: Principal Investigator, Alda Sofia Pires de Dias Marques, Senior Lecturer, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SFRH/BD/148741/2019
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Interstitial Lung Diseases (ILD)
Keywords: Physical activity; Home-based; Interstitial lung diseases; Lifestyle
MeSH Terms: conditions — Lung Diseases, Interstitial; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention model
Who Masked: Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based physical activity group (Experimental): The experimental group will receive the iLiFE.
  Interventions: Other: Home-based physical activity programme
- Control group (Active Comparator): The control group will receive a leaflet with exercises and PA recommendations.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Home-based physical activity programme — iLiFE is a 12-week individualised programme, adapted to the participants' needs and preferences. This programme will be conducted in participants' home and include everyday tasks to train endurance, balance, flexibility and strength. The intervention incudes face-to-face sessions and phone calls. Face-to-face sessions aim to adapt activities to everyday tasks, increase frequency and/or intensity, monitor progress, clarify doubts, motivate higher daily energy expenditure and manage expectations. Phone-calls aim to clarify doubts and to monitor patients' motivation/evolution, following a motivational interview. At the start of the program, the physiotherapist will be present at all sessions, but these face-to-face visits will decrease over time. Patients will also receive a personalised manual (iLiFE manual) with activities to do in their everyday tasks.
  Arms: Home-based physical activity group
Other: Usual care — Participants will receive a leaflet with exercises and PA recommendations.
  Arms: Control group

SUMMARY:
Interstitial lung diseases (ILD) are a highly incapacitating group of chronic respiratory diseases, leading to disabling symptoms and impaired capacity to perform activities of daily living and health-related quality of life (HRQoL). It is known that people with ILD are highly inactive and sedentary, and in a severe stage of the disease, these people spend most of the time at home, increasing dependency on others, and decrease HRQoL. Physical activity is a cost-effective intervention, which increases the HRQoL, exercise capacity and ability to perform activities of daily living in people with chronic respiratory diseases. However, few home-based physical activity programmes are available, especially in people with ILD. Thus, it is urgent to develop innovative models of PA, closer to patients and adjusted to the patients' routines, to engage and change patients' physical activity levels, enhancing HRQoL.

iLiFE might be promising as it focuses on establishing new behaviours, within selected contexts to stimulate home-based PA. Therefore, iLiFE will be developed, implemented and evaluated in people with ILD.

DETAILED DESCRIPTION:
Interstitial lung diseases (ILD) comprise the most highly incapacitating group of chronic respiratory diseases, with significant morbidity and high mortality.

Physical activity (PA) improves HRQoL, exercise capacity and performance of activities of daily living, control the symptoms and prevent the development of further comorbidities in people with chronic respiratory diseases. However, people with ILD are highly inactive and sedentary and, as the disease progresses, these people spend most of time at home and adhere poorly to interventions, which worsens HRQoL, intensifies clinical decline and increases dependency on others.

Home-based PA programmes, integrated in patients' daily routines, may increase PA levels. Lifestyle Integrated Functional Exercise (LiFE) is a home-based PA programme, which integrates training into daily routines. This programme has shown to be effective in healthy older, however its effectiveness in people with a chronic respiratory disease population is unknown.

Therefore, this study will develop and implement a home-based PA programme, based on LiFE, in patients with advanced ILD and assess its impacts on PA levels, HRQoL and other health-related domains.

The PRIMARY AIM of this study is to assess the effects (short- and mid-term) of a home-based PA programme, based on the LiFE programme, on PA levels and HRQoL of patients with ILD, through a randomised controlled trial (RCT).

Secondary aims are to:

1. establish the feasibility of iLiFE and adherence to the intervention;
2. explore the short- and mid-term effects of the iLiFE on the impact of the disease on patients' life, symptoms, exercise tolerance, muscular strength, balance, and emotional status of patients with ILD;
3. assess the cost-benefit of the iLiFE on unscheduled healthcare resources utilisation, length of hospitalisation and number of respiratory infections.

To accomplish these aims, a feasibility study and a RCT will be conducted. iLiFE will be individually tailored to address each person's motivations and capacities, within the home context, to ensure the development and implementation of an innovative home-based PA intervention. Thus, it is expected that iLiFE will improve the PA levels of patients with ILD, enhancing HRQoL. Ultimately, this innovative research will potentially reduce health-care utilisation and costs, and finally, guide clinical and research practice, as well as policy decision makers, at a national and international level.

Task 1: Literature review

To inform the design of the intervention, the investigators will conduct a systematic review on home-based PA interventions in patients with chronic respiratory diseases according to Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA) guidelines.

Task 2: iLiFE-Feasibility study

A mix-methods feasibility study will be conducted to inform the recruitment procedures and components of iLiFE. Sample size will be determined by the qualitative data saturation. The investigators will use a maximum variation strategy to guide recruitment.

Ethical approval will be obtained, and data protection will be ensured by following the European regulation. Eligible patients will be identified by general practitioners or by pulmonologists, who will provide a brief explanation about the study and inform the researcher about interest participants. Then, those interested will be contacted and informed consent obtained. Participants will be eligible if are: i) ≥18 years; ii) diagnosed with stable ILD, in an advanced stage, as determined by referred doctor; iii) living at home. Participants will be excluded if: i) have a history of acute cardiac/respiratory condition on the previous month, and ii) present signs of cognitive impairment or significant cardiovascular, neurological and/or musculoskeletal disease, which may limit participation.

Data will be collected (approximately 1h) at baseline, 4-weeks (after the programme beginning) and 12-weeks (immediately after the programme). The researcher will collect:

* Sociodemographic/anthropometric and general clinical data (e.g., smoking habits, number of exacerbations, healthcare utilisation, and hospitalisation): structured questionnaire;
* PA (steps per day): accelerometry;
* HRQoL: St. George Respiratory Questionnaire;
* Impact of the disease on patients' life: COPD Assessment Test (CAT);
* Dyspnoea: Modified Medical Research Council questionnaire (mMRC) and modified Borg scale;
* Peripheral muscle strength: Handheld dynamometry and handgrip;
* Functional capacity: Time Up and Go test; Brief-Balance Evaluation Systems Test and Physical Performance Test;
* Exercise tolerance: Chester step test;
* Emotional status: Hospital Anxiety and Depression Scale;
* Activities of daily living: London Chest Activity of Daily Living;
* Self-perception of performance in everyday living: The Canadian Occupational Performance Measure (COPM);
* Fatigue: Borg modified scale and Functional Assessment of Chronic Illness Therapy - Fatigue Scale;
* Cough and sputum: Cough and Sputum Assessment questionnaire;
* Occurrence of adverse events and adherence to the interventions.

Accelerometers will be used for 1-week (8h/day) before and after the 12-weeks. The COPM will be used to develop the individualised programme for each patient based on participants' goals.

Individual semi-structured interviews will be conducted, before and after the programme, to inform about patients' preferences, perspectives, barriers and facilitators for programme participation.

iLiFE will be conducted for 12 weeks in participants' homes and will include everyday tasks to train endurance, balance, flexibility and strength. Activities will include: 1) walking and/or stair climbing to improve endurance; 2) functional-based incorporated in activities of daily living, to improve balance (work at the kitchen while standing on one leg), flexibility (stretch the upper limb when watching TV) and muscle strength (squatting instead of bending at the waist to close a drawer or to pick things up from the floor). Intensity of training will be adjusted to perceived exertion confirmed by heart rate and oxygen saturation levels. PA programme will be individualised and based on the results of the assessment.

At the start of the program, the physiotherapist will be present at all sessions, but these face-to-face visits will decrease over time using the following schedule:

* Weeks 1-4: 3 face-to-face sessions/week;
* Weeks 5-8: 2 face-to-face sessions/week and a weekly phone call;
* Weeks 9-11: 1 face-to-face session/week and a weekly phone call;
* Week 12: 2 phone calls.

Face-to-face sessions aim to adapt activities to everyday tasks, increase frequency and/or intensity, monitor progress, clarify doubts, motivate higher daily energy expenditure and manage expectations. Phone-calls aim to clarify doubts and to monitor patients' motivation/evolution, following a motivational interview. Patients will also receive a personalised manual (iLiFE manual) with activities to do in everyday tasks.

Task 3: iLiFE randomised controlled trial

Based on the findings of the literature review and feasibility study, the intervention will be refined.

A sample size calculation was computed for the primary outcome measure (daily steps). Based on a home-based pulmonary rehabilitation study conducted in patients with chronic obstructive pulmonary disease, it is anticipated that 42 participants in each group (total=84) will be needed to detect a between-group difference of 520 steps/day (power=80%, α=0.05, 2-tailed), assuming a strong correlation among paired measures (r=0.70). Since in respiratory interventions dropout rates are around 20%, 100 participants will be needed.

Patients will be randomised into experimental group (EG) and control group (CG). The EG will receive the iLiFE programme described in task 2 and, the CG will receive a leaflet with exercise and PA recommendations.

Data will be collected as described in task 2, however, follow-up assessments will be conducted at 3 and 6 months after iLiFE, to assess short- and mid-term results. In this task, all assessments will be performed by a second researcher blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of a interstitial lung disease
* clinically stable in the previous month
* ≥ 18 years old
* Living at home, assisted-home or at familiar home.

Exclusion Criteria:

* cognitive impairments
* inability to understand and co-operate
* history of neoplasic /immunologic disease or acute cardiac condition or a significant cardiac, musculoskeletal, neuromuscular or psychiatric condition
* Participating in pulmonary rehabilitation or have participated in last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity levels (steps/day) at 12-weeks | Assessment at baseline and 12-week (immediately after iLiFE)
  Accelerometer-based activity monitors. Physical activity levels will be collected with the activity monitors GT3X+ (ActiGraph) to measure the number of steps/day.
Change in Physical activity levels (steps/day) at 3 months | Assessment at baseline and 3 months after iLiFE.
  Accelerometer-based activity monitors. Physical activity levels will be collected with the activity monitors GT3X+ (ActiGraph) to measure the number of steps/day.
Change in Physical activity levels (steps/day) at 6 months | Assessment at baseline and 6 months after iLiFE.
  Accelerometer-based activity monitors. Physical activity levels will be collected with the activity monitors GT3X+ (ActiGraph) to measure the number of steps/day.
Change in physical activity levels (time spent in sedentary, light, lifestyle, moderate and vigorous physical activities) | Multiple time points through study completion - immediately after iLiFE, and up to 3 and 6 months after iLiFE.
  Accelerometer-based activity monitors. Physical activity levels will be collected with the activity monitors GT3X+ (ActiGraph) to measure the daily energy expenditure during one week.

SECONDARY OUTCOMES:
Change in health-related quality of life - The King's Brief Interstitial Lung Disease (KBILD) questionnaire. | Assessment at baseline, 12-week (immediately after iLiFE), 3 and 6 months after iLiFE.
  The King's Brief Interstitial Lung Disease (KBILD) will be used to assess health related quality-of-life. The SGRQ is a comprehensive well-established 50-item questionnaire to measure health status in patients with ILD. Scores can be provided for each domain (symptoms, activities and impact) and as a total score, ranging from 0 (no impairment) to 100 (worst possible health status).
Change in symptom's impact in patients' life | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  COPD Assessment Test (CAT) will be used to assess burdensome symptoms in patients' life with 8 items (cough, sputum, dyspnoea, chest tightness, capacity of exercise and home daily activities, confidence leaving home, sleep and energy levels). The scores range from 0-40, organised in 4 categories, namely <10 low impact, 10-20 medium, 21-30 high and >30 very high impact, with 5 representing the upper limit of normal in healthy non-smokers.
Change in self-reported dyspnoea | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Patients' self-reported level of dyspnoea will be collected at rest, using the modified Borg scale. It is a 10-point scale, rated from 0 to 10, where 0 represents no breathing difficulties, and 10 maximal breathing difficulty.
Change in quadriceps muscle strength | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Quadriceps muscle strength will be measured using a handheld dynamometer (kilogram/force).
Change in handgrip strength | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Handgrip strength will be measured with a dynamometer (kg).
Change in functional status (1-minute sit-to-stand test) | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Participants' functional status will be assessed with the 1-minute sit-to-stand test, which consists in counting the time (seconds) to raise from a chair, walk 3 meters at a comfortable pace, turn, walking back and seat on the chair. Lower time indicates better performance.
Change in exercise tolerance | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Patients' exercise capacity will be assessed using the Chester step test, since it is feasible to apply at patients' home.
Change in emotional state | Assessment at baseline, 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Hospital Anxiety and Depression Scale will be used to assess symptoms of anxiety and depression. It is a 14-item questionnaire that can be subdivided in two subscales: anxiety and depression. Scores are provided for each subscale and range from 0 to 21, with higher scores meaning more symptoms of anxiety and depression.
Change in the impact of breathlessness on activities of daily living | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  London Chest Activity of Daily Living will be used to assess the impact of breathlessness on activities of daily living (ADL). It is a 15-item questionnaire, subdivided in four domains: self-care, domestic, physical and leisure. A sub-total was calculated for each domain and a total score is formed by the sum of the four components' sub-totals, with high scores indicating a greater limitation to ADL.
Change in self-reported fatigue | Assessment at baseline, 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Patients' self-reported level of fatigue will be collected at rest, using the modified Borg scale. It is a 10-point scale, rated from 0 to 10, where 0 represents no fatigue perception, and 10 maximal fatigue perception.
Change in cough and sputum symptoms | Assessment at baseline, 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  The Cough and Sputum Assessment Questionnaire (CASA-Q) will be used to assess cough and sputum symptoms, based on their reported frequency and severity, and their impact on daily activities. It is a 20-item questionnaire containing 4 domains: cough symptoms, cough impact, sputum symptoms and sputum impact. All items are rescored and summed, achieving a score ranging from 0 to 100 for each domain, with higher scores indicating fewer symptoms or less cough and sputum impact.
Change in frequency of exacerbations | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Number of exacerbations in the previous year.
Change in healthcare utilization (number of participants that visits emergency department) | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Healthcare utilization will be assessed through the number of participants that visit emergency department, in the previous year.
Change in functional dyspnoea | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Medical Research Council scale will be used to assess functional dyspnoea related to respiratory impairment. It is a 5-point scale, rated from 0 to 4, with higher scores indicating greater breathlessness severity.
Change in functional status (physical performance test) | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  The physical performance test will be used to assess the overall functionality and evaluates multiple domains of physical function using tasks that simulate activities of daily living. This measure has 9-items with a total score of 36 points, with higher scores indicating better performance.
Change in fatigue | Assessment at baseline, 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  The Functional assessment of chronic illness therapy - fatigue subscale will be used to assess fatigue levels. It is multi-dimensional 13-item questionnaire assessing tiredness, weakness and difficulty in handling daily activities due to fatigue. Scores range from 0 to 52, with higher scores indicating less fatigue.
Change in healthcare utilization (number of visits of each participant) | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Healthcare utilization will be assessed through the number of visits of each participant in the previous year.
Change in healthcare utilization (number of hospital admissions) | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Healthcare utilization will be assessed through the number of hospital admissions in the previous year.
Change in healthcare utilization (duration of hospital admissions) | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Healthcare utilization will be assessed through duration of hospital admissions in the previous year.

OTHER OUTCOMES:
Change in Body Mass Index | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  Patients' body mass index will be assessed in kg/m^2 based on patients' height (in meters) and weight (in kilograms).
Change in number of medications. | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  This outcome will be assessed by the number of medications that each patient takes per day.
Change in the dose of medication | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  This outcome will be assessed by the dose of medication each patient takes per day.
Change in the frequency of medication | Assessment at baseline, 4-weeks (after the programme start), 12-weeks (immediately after iLiFE), 3 and 6 months after iLiFE.
  This outcome will be assessed by the frequency of medication (times/day).

CONTACTS AND LOCATIONS:
Overall Officials: Alda S. Marques, PhD, Principal Investigator — School of Health Sciences of the University of Aveiro (ESSUA)
Locations (1):
- University of Aveiro, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tonelli R, Cocconcelli E, Lanini B, Romagnoli I, Florini F, Castaniere I, Andrisani D, Cerri S, Luppi F, Fantini R, Marchioni A, Beghe B, Gigliotti F, Clini EM. Effectiveness of pulmonary rehabilitation in patients with interstitial lung disease of different etiology: a multicenter prospective study. BMC Pulm Med. 2017 Oct 10;17(1):130. doi: 10.1186/s12890-017-0476-5. PMID 29017478
- [Background] Dowman L, Hill CJ, Holland AE. Pulmonary rehabilitation for interstitial lung disease. Cochrane Database Syst Rev. 2014 Oct 6;(10):CD006322. doi: 10.1002/14651858.CD006322.pub3. PMID 25284270
- [Background] Ryerson CJ, Cayou C, Topp F, Hilling L, Camp PG, Wilcox PG, Khalil N, Collard HR, Garvey C. Pulmonary rehabilitation improves long-term outcomes in interstitial lung disease: a prospective cohort study. Respir Med. 2014 Jan;108(1):203-10. doi: 10.1016/j.rmed.2013.11.016. Epub 2013 Dec 4. PMID 24332409
- [Background] Shah RJ, Collard HR, Morisset J. Burden, resilience and coping in caregivers of patients with interstitial lung disease. Heart Lung. 2018 May-Jun;47(3):264-268. doi: 10.1016/j.hrtlng.2018.03.004. Epub 2018 Apr 4. PMID 29627072
- [Background] World Health Organization. Steps to health: A European framework to promote physical activity for health. Copenhagen: WHO Regional Office for Europe; 2007.
- [Background] Coultas DB, Jackson BE, Russo R, Peoples J, Singh KP, Sloan J, Uhm M, Ashmore JA, Blair SN, Bae S. Home-based Physical Activity Coaching, Physical Activity, and Health Care Utilization in Chronic Obstructive Pulmonary Disease. Chronic Obstructive Pulmonary Disease Self-Management Activation Research Trial Secondary Outcomes. Ann Am Thorac Soc. 2018 Apr;15(4):470-478. doi: 10.1513/AnnalsATS.201704-308OC. PMID 29283670
- [Background] Root ED, Graney B, Baird S, Churney T, Fier K, Korn M, McCormic M, Sprunger D, Vierzba T, Wamboldt FS, Swigris JJ. Physical activity and activity space in patients with pulmonary fibrosis not prescribed supplemental oxygen. BMC Pulm Med. 2017 Nov 23;17(1):154. doi: 10.1186/s12890-017-0495-2. PMID 29169394
- [Background] Perez-Bogerd S, Wuyts W, Barbier V, Demeyer H, Van Muylem A, Janssens W, Troosters T. Short and long-term effects of pulmonary rehabilitation in interstitial lung diseases: a randomised controlled trial. Respir Res. 2018 Sep 20;19(1):182. doi: 10.1186/s12931-018-0884-y. PMID 30236104
- [Background] Wickerson L, Mathur S, Helm D, Singer L, Brooks D. Physical activity profile of lung transplant candidates with interstitial lung disease. J Cardiopulm Rehabil Prev. 2013 Mar-Apr;33(2):106-12. doi: 10.1097/HCR.0b013e3182839293. PMID 23403914
- [Background] Interventions on Diet and Physical Activity: What Works: Summary Report. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK177205/ PMID 24432437
- [Background] Clemson L, Fiatarone Singh MA, Bundy A, Cumming RG, Manollaras K, O'Loughlin P, Black D. Integration of balance and strength training into daily life activity to reduce rate of falls in older people (the LiFE study): randomised parallel trial. BMJ. 2012 Aug 7;345:e4547. doi: 10.1136/bmj.e4547. PMID 22872695
- [Background] • World Health Organization. International Classification of Functioning, Disability and Health. ICF checklist. 2001.
- [Background] Holland AE, Mahal A, Hill CJ, Lee AL, Burge AT, Cox NS, Moore R, Nicolson C, O'Halloran P, Lahham A, Gillies R, McDonald CF. Home-based rehabilitation for COPD using minimal resources: a randomised, controlled equivalence trial. Thorax. 2017 Jan;72(1):57-65. doi: 10.1136/thoraxjnl-2016-208514. Epub 2016 Sep 26. PMID 27672116
- [Background] Borg G. Borg's perceived exertion and pain scales. HUman kinetics. 1998.
- [Background] Papiris SA, Daniil ZD, Malagari K, Kapotsis GE, Sotiropoulou C, Milic-Emili J, Roussos C. The Medical Research Council dyspnea scale in the estimation of disease severity in idiopathic pulmonary fibrosis. Respir Med. 2005 Jun;99(6):755-61. doi: 10.1016/j.rmed.2004.10.018. Epub 2004 Nov 24. PMID 15878493
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Graham BL, Brusasco V, Burgos F, Cooper BG, Jensen R, Kendrick A, MacIntyre NR, Thompson BR, Wanger J. Executive Summary: 2017 ERS/ATS standards for single-breath carbon monoxide uptake in the lung. Eur Respir J. 2017 Jan 3;49(1):16E0016. doi: 10.1183/13993003.E0016-2016. Print 2017 Jan. PMID 28049167
- [Background] Spruit MA, Sillen MJ, Groenen MT, Wouters EF, Franssen FM. New normative values for handgrip strength: results from the UK Biobank. J Am Med Dir Assoc. 2013 Oct;14(10):775.e5-11. doi: 10.1016/j.jamda.2013.06.013. Epub 2013 Aug 16. PMID 23958225
- [Background] Dowman L, McDonald CF, Hill CJ, Lee A, Barker K, Boote C, Glaspole I, Goh N, Southcott A, Burge A, Ndongo R, Martin A, Holland AE. Reliability of the hand held dynamometer in measuring muscle strength in people with interstitial lung disease. Physiotherapy. 2016 Sep;102(3):249-55. doi: 10.1016/j.physio.2015.10.002. Epub 2015 Oct 22. PMID 26596172
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] • Guralnik JM. Assessing Physical Performance in the Older Patient [CD-ROM]. In: Bethesda MD: National Institutes of Aging, editor. 2013.
- [Background] Reuben DB, Siu AL. An objective measure of physical function of elderly outpatients. The Physical Performance Test. J Am Geriatr Soc. 1990 Oct;38(10):1105-12. doi: 10.1111/j.1532-5415.1990.tb01373.x. PMID 2229864
- [Background] Skyes K. Chester Step Test. Publications WA, editor2003.
- [Background] Direção-Geral da Saúde. Diagnóstico e tratamento da doença pulmonar obstrutiva crónica: norma nº 028/2011, de 30/09/2011, atualização de 10/09/2013. DGS Lisboa; 2013.
- [Background] Reilly CC, Bausewein C, Garrod R, Jolley CJ, Moxham J, Higginson IJ. Breathlessness during daily activity: The psychometric properties of the London Chest Activity of Daily Living Scale in patients with advanced disease and refractory breathlessness. Palliat Med. 2017 Oct;31(9):868-875. doi: 10.1177/0269216316680314. Epub 2016 Dec 15. PMID 27932629
- [Background] Pitta F, Probst VS, Kovelis D, Segretti NO, Mt Leoni A, Garrod R, Brunetto AF. Validation of the Portuguese version of the London Chest Activity of Daily Living Scale (LCADL) in chronic obstructive pulmonary disease patients. Rev Port Pneumol. 2008 Jan-Feb;14(1):27-47. English, Portuguese. PMID 18265916
- [Background] Pais-Ribeiro J, Silva I, Ferreira T, Martins A, Meneses R, Baltar M. Validation study of a Portuguese version of the Hospital Anxiety and Depression Scale. Psychol Health Med. 2007 Mar;12(2):225-35; quiz 235-7. doi: 10.1080/13548500500524088. English, Portuguese. PMID 17365902
- [Background] Webster K, Cella D, Yost K. The Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System: properties, applications, and interpretation. Health Qual Life Outcomes. 2003 Dec 16;1:79. doi: 10.1186/1477-7525-1-79. PMID 14678568
- [Background] Gries KS, Esser D, Wiklund I. Content validity of CASA-Q cough domains and UCSD-SOBQ for use in patients with Idiopathic Pulmonary Fibrosis. Glob J Health Sci. 2013 Sep 16;5(6):131-41. doi: 10.5539/gjhs.v5n6p131. PMID 24171881
- [Background] Swigris JJ, Esser D, Wilson H, Conoscenti CS, Schmidt H, Stansen W, Leidy NK, Brown KK. Psychometric properties of the St George's Respiratory Questionnaire in patients with idiopathic pulmonary fibrosis. Eur Respir J. 2017 Jan 18;49(1):1601788. doi: 10.1183/13993003.01788-2016. Print 2017 Jan. PMID 28100551
- [Background] Dedding C, Cardol M, Eyssen IC, Dekker J, Beelen A. Validity of the Canadian Occupational Performance Measure: a client-centred outcome measurement. Clin Rehabil. 2004 Sep;18(6):660-7. doi: 10.1191/0269215504cr746oa. PMID 15473118
- [Background] Holland AE, Watson A, Glaspole I. Comprehensive pulmonary rehabilitation for interstitial lung disease: A consensus approach to identify core education topics. Patient Educ Couns. 2019 Jun;102(6):1125-1130. doi: 10.1016/j.pec.2019.01.010. Epub 2019 Jan 16. PMID 30683609